CLINICAL TRIAL: NCT00778882
Title: An Open-label, Uncontrolled, Single Center, Phase I/II Trial to Assess the Safety and Efficacy of Autologous Hematopoietic Stem Cells Transduced With MT-gp91 Retroviral Vector in gp91 Defective Chronic Granulomatous Disease Patients
Brief Title: Gene Therapy for Chronic Granulomatous Disease in Korea
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This Korean Phase 1 study was Withdrawn more than 15 years ago and no data is available.
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VM106-KR-01
Record Dates: First submitted 2008-10-21; First posted 2008-10-24 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Chronic Granulomatous Disease
Keywords: Chronic Granulomatous Disease; Retroviral Vector; Gene Therapy
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VM106 (Experimental)
  Interventions: Drug: VM106

INTERVENTIONS:
Drug: VM106 — Autologous hematopoietic stem cells with MT-gp91 retroviral vector

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of administration of autologous hematopoietic stem cells transduced with MT-gp91 retroviral vector for patients with X-linked chronic granulomatous disease.

ELIGIBILITY:
Inclusion Criteria:

* gp91 defective male patients with chronic granulomatous disease: confirmed by DHR
* Weigh greater than or equal to 15 kg
* History of severe infections: more than 2 times
* Performance status: ECOG 0-2
* Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

  * Heart: a shortening fraction > 28%; QTc interval < 0.44
  * Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal; AST < 3 x upper limit of normal
  * Kidney: creatine < 2 x normal
  * Blood: WBC > 2,500/uL; platelet > 100,000/uL; hematocrit > 26%
* Written informed consent obtained from patient (or guardian if patients age < 19)

Exclusion Criteria:

* Presence of a HLA-matched sibling for stem cell donation
* Evidence or history of malignant tumor
* Presence of a severe infection
* Presence of an active tuberculosis
* Uncorrectable electrolyte, Ca, P
* Unable to comply with the protocol or to cooperate fully with the Investigator or site personnel

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01 (Estimated); Primary Completion 2008-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events through 1 year | 1 year

SECONDARY OUTCOMES:
RCR, insertional mutagenesis, immune response against normal gp91 protein | 1 year
Safety and efficacy of fludarabine/busulfan conditioning | 1 year
Functional reconstitution of respiratory burst | 1 year
Presence of vector-positive cells | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joong Gon Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea